CLINICAL TRIAL: NCT05474521
Title: Evaluation of Illinois Agility Performance With Smartphone Applications: A Validity and Reliability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Huseyin Sahin UYSAL, Research Assistant, Mehmet Akif Ersoy University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: MehmetAkifU
Record Dates: First submitted 2022-07-20; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Training Group; Sensitivity
Keywords: Performance test; Smarthone app; Agility
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: This study was performed according to the predictive correlational research design, which is one of the quantitative research methods. Participants included in the study were determined according to the simple random sampling method. Athletes who studied at the faculty of sports sciences participated in this research and the research was carried out with a single group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (30):
- Participant 1 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 2 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 3 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 4 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 5 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 6 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 7 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 8 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 9 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 10 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 11 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 12 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 13 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 14 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 15 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 16 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 17 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 18 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 19 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 20 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 21 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 22 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 23 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 24 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 25 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 26 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 27 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 28 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 29 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test
- Participant 30 (Experimental): The participant applied the Illinois test twice to determine the validity, reliability, and usefulness of the data collection tools.
  Interventions: Device: CODTimer test

INTERVENTIONS:
Device: CODTimer test — The Illinois test times of the participants will be measured with different phone applications that measure the change of direction performance, and each individual will perform the test twice.
  Other Names: Stopwatch Moviewatch App; Seconds Count; Stopwatch; Photocell

SUMMARY:
Due to the impracticality of accessing the gold standard test devices, researchers have developed easy-to-use and cost-effective smartphone applications that do not require expert knowledge, and these applications have been used to measure different motor abilities. Smartphone applications such as CODtimer, Stopwatch Movie watch, and Seconds Count are used to evaluate the ability to change direction within these biomotor features. However, the validity and reliability of these applications are the subjects of research.

DETAILED DESCRIPTION:
The athletic performance level is one of the main factors that determine the success of an athlete. However, the athletic performance level of an athlete is determined by many motor abilities. One of these motor abilities is agility.

Because agility has been seen as a complex physical skill, valid and reliable tests and test devices are needed to determine the level of agility. Therefore, researchers have developed many test devices using technology and they have aimed to reach gold standards to measure agility ability through these devices. In this context, manual timers were first used to measure agility performance, then devices such as fully automatic test devices, photocell types, video timers, and radar systems were accepted as a test tool for the measurement of agility performance. Although fully automatic test devices are accepted as the gold standard in the measurement of velocity-based parameters, they cannot be preferred by everyone due to obstacles such as the need for expert knowledge and being economically costly for their use.

Due to the impracticality of accessing the gold standard test devices, researchers have developed easy-to-use and cost-effective smartphone applications that do not require expert knowledge, and these applications have been used to measure different motor abilities. Among these motor features, CODTimer App is the smartphone application that is frequently preferred in the evaluation of agility ability and whose validity-reliability studies are conducted.

In the previous studies on the validity and reliability of the CODTimer App, a very strong correlation was found between the CODTimer App and the gold standard automatic timing gates according to the 5+5 and 505 agility test protocols. However, many mobile applications have validity and reliability unexplored. It is necessary to investigate different test protocols and devices to spread the use of mobile applications and prove that they are valid and reliable measurement tools.

This study aimed to determine the validity, reliability, and usefulness of the CODTimer, Second Count, and Stopwatch Moviewatch App with an iPhone 11 compared to gold standard timing gates for the evaluation of Illinois agility performance in college athletes.

ELIGIBILITY:
Inclusion Criteria:

* Athletes who have not experienced an injury in the last 1 year and have a training history of at least one year.

Exclusion Criteria:

* Participants who do not meet the inclusion criteria

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
The relationship of smartphone apps versus gold standard measuring tool in measuring direction change performance | 1-week
  Two photocell doors with a height of 1.5 meters and a distance of 2 meters were placed at the beginning and the end of the test. However, to take measurements with smartphone applications, video recordings were made with smartphones from a height of 1.5, 2 meters away from the photocell, parallel to the ending and starting points. To measure with the stopwatch, the researchers were positioned 1 meter next to the photocell at the endpoint. At the beginning of the test, the exit positions of the participants were standardized, and each participant applied the illinois test twice with three minutes of listening.
  The means of the obtained values were determined according to the following formula; (first trial time[second]+ second trial time[second])/2. Hypothesis tests were performed with trial time mean. It was assumed that the shorter the test times of the athletes, the better their performance.

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin Sahin Uysal, Msc, Study Director — Burdur Mehmet Akif Ersoy University
Locations (2):
- Turkey (Türkiye) (2):
  - Burdur Mehmet Akif Ersoy University Faculty of Sport Science, Burdur
  - Huseyin Sahin UYSAL, Burdur

IPD SHARING:
Plan to Share IPD: Undecided